CLINICAL TRIAL: NCT06954922
Title: The Effect of Memory-Based Exercise and Planned Training Applied to Epilepsy Patients on Quality of Life
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, AHMET ŞİMŞEK, PhD student, Ataturk University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: ATAÜNİ-SBE-AS-02
Record Dates: First submitted 2025-04-10; First posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Epilepsy; Memory Consolidation; Education of Patients; Quality of Life (QOL)
Keywords: quality of life; epilepsy; education of patiens; memory
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- memory-based exercise and training group (Experimental)
  Interventions: Behavioral: memory-based exercise and training intervention
- training group (Experimental)
  Interventions: Behavioral: educational initiative about epilepsy

INTERVENTIONS:
Behavioral: memory-based exercise and training intervention — The experimental group will be given memory-based exercises that will last approximately 15-20 minutes every day for 2 months. Four sessions of epilepsy training will be given, one session per week.
  Arms: memory-based exercise and training group
Behavioral: educational initiative about epilepsy — This group will be given 4 sessions of epilepsy training, one session per week.
  Arms: training group

SUMMARY:
Epilepsy; It is a chronic, neurological disease that can occur regardless of social class, race and age. Every year, approximately 5 million people worldwide are diagnosed with epilepsy and 50 million people are affected by this disease, constituting a significant part of the disease burden in the world. When we look at the rate of patients in the population who actively experience symptoms of the disease and need treatment, this rate is approximately 4 to 10 people per 1000 people. According to estimates, 700,000 people in Turkey are actively diagnosed with epilepsy. It is accepted that this disease occurs as a result of sudden, abnormal discharge of neurons in some parts of the central nervous system, and the disease generally progresses with recurrent changes in consciousness. The symptoms accompanying epilepsy are perceived negatively by patients and significantly affect their lives. Epilepsy treatment; It consists of several options such as medical drugs, ketogenic diet and surgical intervention. The ultimate goal of treatment is to achieve seizure control, reduce the frequency of seizures, minimize drug side effects that may occur due to long-term treatment, and improve the patient's quality of life. Along with pharmacological treatment, non-pharmacological treatment is also a valuable approach in the treatment of epilepsy. One of the non-pharmacological approaches is rehabilitation interventions with mind and memory exercises. Epilepsy is a disease that requires a complex psychological adaptation for the patient and affects the whole family. In this disease, it is very important for the patient to comply with the treatment requirements, to have self-control over his/her behavior, as well as to cope with the difficulties of living with epilepsy. Increasing the quality of life and preventing possible behavioral problems is possible by keeping mental functions at an optimal level on the one hand, and providing psychological counseling to the patient and his family on the other. Nowadays, epileptic seizures are often more easily controlled with developing pharmacological treatment options. Therefore, the fight against epilepsy should be expanded to include other educational, mental, psychotherapeutic and behavioral interventions besides drug therapy. In a study conducted by the National Center for Health and Care Research (NIHR), electrical activity scans in the brain of 25 epilepsy patients were examined. Some images in different categories were presented to epilepsy patients for a certain period of time. Later, when asked to remember the images shown in the previous step, it was noted that slow waves occurred in the brain during sleep. As a result of the research, it was revealed that the effect of epileptic spikes on brain activity decreased with the emergence of slow waves. This study has demonstrated for the first time a potential protective mechanism used by the brain to counteract epileptic activity. Patients diagnosed with epilepsy who are admitted to the neurology outpatient clinic or admitted to the neurology clinic will be introduced and informed about the study. Patients who want to participate in the study and meet the inclusion criteria will be determined. After patient consent is obtained, groups will be determined according to the randomization list.

The patient introduction form and the Quality of Life in Epilepsy Scale will be administered to the patients in both groups by the researcher using the face-to-face interview technique (pre-test). Patients in the experimental group will be informed about memory-based exercise and planned training.

Patients in the control group will only be informed about the planned training to be given.

The experimental group will be given memory-based exercises that will last approximately 15-20 minutes every day for 2 months. Four sessions of epilepsy training will be given, one session per week.

The control group will receive 4 sessions of epilepsy training, one session per week.

At the end of two months, the Quality of Life in Epilepsy Scale (posttest) will be applied to both groups.

ELIGIBILITY:
Inclusion Criteria:

1. Being literate,
2. Being over the age of 18,
3. Having sufficient communication skills to answer oral and written questions and follow instructions,
4. Being at a cognitive level to be able to use a mobile phone and perform the memory exercise.
5. Not having severe vision problems,
6. Having been diagnosed with epilepsy for at least 6 months

Exclusion Criteria:

1. Being under 18 years of age
2. Residing outside Bilecik Province
3. Having psychiatric diagnoses such as Bipolar Disorder and Schizophrenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Patient Introduction Form | 2 month
  It was prepared by the researcher by examining the literature. It consists of 26 questions, including questions such as age, gender, marital status, educational status, family type, social security, income status, epilepsy diagnosis period, frequency of seizures, presence of another disease, constantly used medication.
Quality of Life Scale in Epilepsy | 2 month
  QOLIE-31 was developed by Vickrey et al. in 1993. Mollaoğlu and his colleagues were the researchers who conducted the validity and reliability studies of this scale in Turkey in 2015. QOLIE-31; It consists of a total of 31 questions and 7 subcomponents: 5 on the seizure-related concerns sub-dimension, 3 on the effects of medications sub-dimension, 4 on the energy/fatigue sub-dimension, 5 on the emotional well-being sub-dimension, 6 on the cognitive function sub-dimension, 5 on the social function sub-dimension, 2 on the total quality of life sub-dimension and an additional question assessing the total health status. Scale scoring ranges from 0-100 points. A high score indicates a high quality of life. The total Cronbach's Alpha value in the original scale was determined to be 0.91. In this study, the total Cronbach Alpha value of the scale was found to be 0.90.